CLINICAL TRIAL: NCT06691529
Title: The Association of Metabolic Associated Fatty Liver Disease in Patients With Chronic Glomerular Disease
Brief Title: Metabolic Associated Fatty Liver Disease in Patients With Chronic Glomerular Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Samar Fahmy Amin Sayed, physician, Assiut University
Other Study IDs: fatty liver disease
Record Dates: First submitted 2024-11-14; First posted 2024-11-15 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Fatty Liver Disease; Chronic Glomerular Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: 500 patients presented at Nephrology unit/Internal Medicine department (Assiut University Hospital) In the period 2024-2026.

SUMMARY:
The association of metabolic associated fatty liver disease in patients with chronic glomerular disease

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is associated with high morbidity and mortality, and is rapidly becoming a major burden to the global health care system.

Chronic kidney disease CKD is a complex, progressive chronic condition that is defined by either abnormality of kidney structure or function present for ≥3 months Either markers of kidney damage or decreased glomerular filtration rate may be present.

The global prevalence of CKD was estimated at 10.4-13.4% , stage 5 HD is rapidly increasing worldwide and expected to further increase in the next decade .

Metabolic associated fatty liver disease (MAFLD) is characterized by excessive hepatic fat accumulation without significant alcohol intake, use of medications causing fatty liver, or other traditional causes of fatty liver, is the most common cause of chronic liver disease worldwide, especially in developed countries . MFLD refers to a wide spectrum of liver damage, ranging from simple steatosis to non-alcoholic steatohepatitis, advanced fibrosis and cirrhosis Studies have shown that MAFLD is the underlying cause of an increasing number of extrahepatic manifestations. MAFLD is mainly linked to type II diabetes mellitus (T2DM) and cardiovascular disease (CVD), as well as a number of other severe chronic diseases including chronic kidney disease (CKD) The diagnosis of MAFLD requires the presence of hepatic steatosis plus at least one of the following three metabolic risk abnormalities: overweight/obesity, T2DM or evidence of metabolic dysregulation.

Metabolic syndrome (MetS) was defined according to the National Cholesterol Education Program ATP III criteria (16) as the presence of any three or more of the following metabolic conditions: Abdominal obesity, waist circumference ⩾ 102 cm in men and ⩾ 88 cm in women. Serum triglycerides (TG) ⩾ 150 mg/dL (1.7 mmol/L) or drug treatment for elevated triglycerides, serum high-density lipoprotein cholesterol<40 mg/dL (1.0 mmol/L) in men and<50 mg/dL (1.3 mmol/L) in women or drug treatment for low high density lipoprotein cholesterol. Blood pressure ⩾ 130/85 mmHg or drug treatment for elevated blood pressure, fasting blood glucose ⩾ 100 mg/dL (5.6 mmol/L) or drug treatment for elevated blood glucose.

Diabetes mellitus (DM) was defned as a fasting blood glucose level of ⩾125 mg/dl, or prescription of antidiabetic drugs, Hypertension was defned as systolic blood pressure (SBP) ⩾ 130 mmHg, diastolic blood pressure (DBP) ⩾ 85 mmg , or prescription of antihypertensive drugs.

A recent meta-analysis of about 10 million individuals reported a global prevalence of MAFLD of 38.8% in adults. In addition, it has been reported that MAFLD may progress to cirrhosis and promote the development of some important extrahepatic diseases, such as cardiovascular disease and chronic kidney disease (CKD).

MAFLD and CKD share some common features, including visceral obesity, T2DM, hypertension and metabolic syndrome and both diseases are also linked to an increased risk of CVD . Both diseases are progressive chronic conditions that represent a spectrum of diseases extending from relatively mild disease, with only modest changes in function, to severe debilitating disease with end-stage organ damage, necessitating either chronic dialysis or organ transplantation in order to sustain life.

The potential relationship between NAFLD and CKD has recently attracted scientists' interest. Establishing a relationship between liver and kidney injury would help to identify kidney illness sooner and enable for the selection of medicines that target both liver and kidney disease, with potentially beneficial preventative and therapeutic implications .

ELIGIBILITY:
Inclusion Criteria:

* All CKD patient aging between (18-70) years with known tubule-glomerular diseases.
* At any eGFR.
* All CKD patient have either type I/II DM associated with CKD .

Exclusion Criteria:

* CKD patients of Unknown etiology.
* CKD patients with liver cirrhosis.
* CKD patients secondry to documented diabetic nephropathy.
* Patients with previous/current HBV or HCV.
* Pregnant CKD patients.
* Patient commencing any hepatotoxic medication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in this study will be subjected to
  1. Detailed history and full clinical examination
  2. Anthropometric measurements; Hight, weight, waist circumference.
  3. Full lab investigations (Complete blood picture , kidney function tests, liver function tests, serum electrolytes, Ferritin, Uric acid level, Prothrombin time and concentration and serum albumin)
  4. High sensitivity CRP
  5. lipid profile (Fasting)
  6. urine analysis, ACR.
  7. Available documented renal biopsy
  8. HBA1c
  9. C- peptide levels. 10. FIB4 - score
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
association between metabolic associated fatty liver disease and chronic kidney disease | through study completion, an average of 1 year
  To detect the association between metabolic associated fatty liver disease and chronic kidney disease with glomerular diseaese in Assuit university hospital.